CLINICAL TRIAL: NCT01865266
Title: The Effect of Ulinastatin on Bronchoalveolar Lavage Fluid of Inflammatory Factors in Patients With Ventilator-associated Pneumonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minhang Central Hospital (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yu YueTian, Shanghai Minhang Central Hospital, Shanghai Minhang Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAP-YYT-003
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Ventilator-associated Bacterial Pneumonia; Mechanical Ventilation Complication
Keywords: ventilator-associated pneumonia; mechanical ventilation; ulinastatin for injection; bronchoalveolar lavage fluid; inflammatory factors
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NUTIG (Experimental): The normal dose of ulinastatin for injection group(NUTIG):
  Ulinastatin(Techpool inc,Guangdong,China) was administered to the group as a bolus of 100,000 U diluted in 100 mL of normal saline every 8 hour.A course of treatment consisted of 7 days after the patients were diagnosed as VAP.
  Interventions: Drug: Ulinaststin for injection
- HUTIG (Experimental): The high dose of ulinastatin for injection group(HUTIG):
  Ulinastatin(Techpool inc,Guangdong,China) was administered to the group as a bolus of 200,000 U diluted in 100 mL of normal saline every 8 hour.A course of treatment consisted of 7 days after the patients were diagnosed as VAP.
  Interventions: Drug: Ulinaststin for injection
- CG (Placebo Comparator): The compare group(CG):
  The group was given 100 mL of normal saline every 8 hour.A course of treatment consisted of 7 days after the patients were diagnosed as VAP.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ulinaststin for injection
  Arms: HUTIG; NUTIG
Drug: placebo
  Arms: CG

SUMMARY:
Ventilator-associated pneumonia (VAP) is an important cause of morbidity and mortality in ventilated critically ill patients specially in intensive care unit (ICU). It is associated with an increased duration of mechanical ventilation, high death rates and increased healthcare costs in the development country.

Although VAP is preventable and many practices have been demonstrated to reduce the incidence of this disease, the morbidity is still so high. VAP is hard to cure and the mortality is about to 40% which was reported in China in 2004. If the bacteria of multidrug-resistance(MDR) is isolated, the mortality can increase to 70%. So much more methods should be needed in treating VAP in addition to using antibiotics.

Ulinastatin is a serine protease inhibitor with a molecular weight of 67,000 found in healthy human urine. It is used worldwide for patients with inflammatory disorders, including disseminated intravascular coagulation(DIC),shock, and pancreatitis . Furthermore, ulinastatin administration can help reduce sepsis, prevent multiple organ dysfunction, and modulate immune functions.

Actually, three studies have showed that ulinastatin treatment is associated with reduced the levels of inflammatory factors in blood serum in patients with acute respiratory distress syndrome(ARDS).Though analyses of serum inflammatory factors such as tumor necrosis factor (TNF)-α and interleukin (IL)-6 have been used to determine the degree of systemic inflammation under various clinical conditions, they can not reflect the degrees of lung infection directly.

Basing on the results of previous studies, meta analyses and system reviews, the investigators hypothesized that the anti-inflammatory function of ulinaststin may also decrease the levels of inflammatory factors in bronchoalveolar lavage(BAL) fluid in Patients with VAP.

In addition there is no prospective study to investigate the role of ulinastatin in BAL. The investigator hopes that this study can approve the relationship between ulinastatin and inflammatory factors in BAL. And it can improve the processes,outcomes and costs of critical care as well.

DETAILED DESCRIPTION:
This is a one-center, three-arm, randomized, single-blinded, controlled trial. When a patient was diagnosed VAP during mechanic ventilation in ICU,a sealed envelop will be opened which decide whether the patient is assigned to the normal dose ulinastatin group,the high dose ulinastatin group or the compare group.

VAP diagnosis and treatment accord with the "Comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia:Diagnosis and treatment" which was published in 2008 by Canadian critical care trials group.

The aim of the present study is to determine the efficacy of ulinastatin for the treatment of ventilator-associated Pneumonia(VAP) and to investigate the effect to inflammatory factors in bronchoalveolar lavage fluid .

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with ventilator-associated pneumonia(VAP) who are admitted to the intensive care unit between 1st January 2014 at 0:00(midnight) and the finish date of 31st December 2015 at 23:59 (11:59 pm).
* Informed consent.

Exclusion Criteria:

* Patients with pneumonia when they are admitted to ICU.
* Ulinastatin was previous used before the patients were diagnosed VAP.
* Active gastropathic disorder.
* Be allergic to ulinastatin.
* Pregnancy.
* Unwilling to continue the therapy during hospitalization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Levels of inflammatory factors in bronchoalveolar lavage fluid and blood serum. | 7 days
  The variety of tumor necrosis factor-α(TNF-α),interleukin-10(IL-10),interleukin-18(IL-18) and interferon-γ(INF-γ) in bronchoalveolar lavage fluid and blood serum are observed.

SECONDARY OUTCOMES:
All cause mortality. | 30 days
Ventilation free days. | 30 days
Antibiotic free days. | 30 days
Percentage of MDR pathogenic bacteria. | 30 days
  We will find whether the bacteria of multidrug-resistance can be isolated from the bronchoalveolar lavage fluid culture.
  We will count the number of methicillin-resistant staphylococcus aureus(MRSA),extended-spectrum beta-lactamase(ESBLs) or vancomycin-resistant enterococcus(VRE) isolated from bronchoalveolar lavage fluid culture.
Oxygenation index | 30 days
  Oxygenation index = Fio2/PaO2(mmHg)

OTHER OUTCOMES:
Adverse effects | 30 days
  The adverse effects from using ulinastatin. Irritability,nausea,vomit,diarrhoea or the aspartate transaminaseere and alanine transaminase are more than one time the upper normal limit were regarded as the adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Minhang Central Hospital, Shanghai, China